CLINICAL TRIAL: NCT05416177
Title: Assessment of Vivity With French Clinical Data Related to the Toric Model Study
Acronym: VICTOR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Edouard KOCH, Investigator Coordinator, Versailles Hospital
Other Study IDs: P21/21 - VICTOR
Record Dates: First submitted 2022-06-03; First posted 2022-06-13 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Presbyopia-correcting implant (PC-IOL): AcrySof IQ Vivity (Alcon) has been evaluated in 2 large pivotal trials (US and OUS trials). These tests showed that this PC-IOL restored intermediate visual acuity (IVA) and near visual acuity (NV A) superior to that of the reference monofocal AcrySof implant. In these tests, it was demonstrated that distance visual acuity (DVA) was non-inferior. However, the intermediate visual acuity for this implant in its toric version has not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for a request for cataract surgery in current practice: phacoemulsification followed by classic implantation of an IOL with small incision size (< 2.2mm)
* Calculated power of IOL is between 10.0 and 30.0 diopters (D) in 0.5D steps to target emmetropia (0.0 +/- 0.5D)
* Patients with corneal astigmatism > 0.5D and who can receive an implant with a toricity between T2 and T6, i.e. with astigmatism between +0.5D and +2.5D.
* If both eyes have astigmatism, the eye under study will be the right eye
* Patient having been informed and not objecting to their participation.

Exclusion Criteria:

* Pregnancy or breastfeeding while conducting the study
* Person under the age of 18
* History of pathologies of the anterior segment of the eye (cornea, anterior chamber, sulcus) or posterior segment of the eye (uvea, vitreous, retina) including retinal vascular occlusions, retinal detachment, peripheral retinal laser photocoagulation, AMD and glaucoma
* Any inflammation of the anterior or posterior segment, whatever its etiology or history of disease, which may lead to an inflammatory reaction
* Clinically significant corneal pathology (epithelial, stromal, or endothelial that could affect visual outcome)
* Clinically significant severe dry eye disease that may affect visual calculations and measurements
* History of refractive surgery
* Amblyopia or monofixation syndrome
* Patient at risk of zonular rupture during the phacoemulsification procedure and may affect the centering or tilt of the implant postoperatively.
* Irregular astigmatism (corneal topography)
* Any other planned eye surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from among patients who come for consultation for cataract surgery. During the inclusion visit, the doctor will inform the patients eligible for the study, and answer all their questions about the objective, the constraints, the foreseeable risks and the expected benefits of the study. Without opposition from the patient, the doctor will perform the cataract surgery and the data will be collected on D0, M1 and M3.
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Distance corrected intermediate monocular visual acuity | month 3
  Intermediate monocular visual acuity (at 66 cm) corrected for distance vision (DCIVA) for the eye under study in photopic condition (normal lighting) 3 months after implantation of the 2nd eye

SECONDARY OUTCOMES:
rotational stability | month 3
  Rotational stability of the IOL in the eye under study expressed in degree of rotation at 3 months compared with that collected just after surgery in the operating room
residual astigmatism | months 1 and 3
  measure of total residual astigmatism including corneal and internal astigmatism in dioptries
monocular distance visual acuity | months 1 and 3
  Corrected (BCDVA) and uncorrected monocular distance visual acuity (UCDVA) for the study eye (at 4 m)
monocular near visual acuity | months 1 and 3
  Corrected (DCNVA) and uncorrected monocular (UCNVA) near visual acuity for the study eye (at 40 cm)
monocular uncorrected intermediate visual acuity | months 1 and 3
  Uncorrected intermediate visual acuity monocular (UCIVA) for the eye under study (at 66 cm)
binocular uncorrected visual acuity | months 1 and 3
  Binocular uncorrected visual acuity (UCVA) from far to 4 m, intermediate at 66 cm, near at 40 cm.
SIA | month 3
  Surgically induced astigmatism (SIA) and comparison between the 2 hospitals participating in the study
questionnaire IOLSAT | month 3
  questionnaire for addiction to glasses for intermediate vision and near vision (IOLSAT) : minimum 0% (no glasses needed, best outcome), to maximum 100% (glasses needed, worse outcome)
McAlinden questionnaire | month 3
  questionnaire for the evaluation of visual disturbances (McAlinden): minimum 0/90 and maximum 90/90 (worse outcome)